CLINICAL TRIAL: NCT07268495
Title: The Impact of Intraperitoneal Spray Combined With Intravenous Lidocaine on Postoperative Pain After Myomectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Shaoling Ma-2025-05
Record Dates: First submitted 2025-08-21; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain
Keywords: lidocaine; myomectomy; laparoscopic surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride; Analgesics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group C(Control Group) (Active Comparator): At the beginning of the operation, intravenous infusion of reifentanil 0.1~0.2μg/kg/min, propofol 2~4mg/kg/h, rocuronium 0.3mg/kg/h intermittently, inhalation of 1%~2% sevoflurane were maintained, the fluctuation of blood pressure was not more than 20% of the basic level, and the heart rate was 50~100 times /min. 10 minutes before the infusion proper amount of normal saline was administered to the patient. Subsequnetly, a continuous intravenous infusion proper amount of normal saline was maintained until the end of the sugery. Before closing the abdominal cavity, 20ml normal saline was administered.
  Interventions: Drug: Saline
- Group IV(Intravenous injection of lidocaine Group) (Experimental): At the beginning of the operation, intravenous infusion of reifentanil 0.1~0.2μg/kg/min, propofol 2~4mg/kg/h, rocuronium 0.3mg/kg/h intermittently, inhalation of 1%~2% sevoflurane were maintained, the fluctuation of blood pressure was not more than 20% of the basic level, and the heart rate was 50~100 times /min. 10 minutes before the infusion 2% lidocaine (1.5mg/kg) was administered to the patient. Subsequnetly, a continuous intravenous 2% lidocaine (2mg/kg/h) was maintained until the end of the sugery. Before closing the abdominal cavity, 20ml normal saline was administered.
  Interventions: Drug: intravenous +saline lidocaine
- Group IP(Intraperitoneal spray of lidocaine Group) (Experimental): At the beginning of the operation, intravenous infusion of reifentanil 0.1~0.2μg/kg/min, propofol 2~4mg/kg/h, rocuronium 0.3mg/kg/h intermittently, inhalation of 1%~2% sevoflurane were maintained, the fluctuation of blood pressure was not more than 20% of the basic level, and the heart rate was 50~100 times /min. 10 minutes before the infusion proper amount of normal saline was administered to the patient. Subsequnetly, a continuous intravenous infusion proper amount of normal saline was maintained until the end of the sugery. Before closing the abdominal cavity, 2% lidocaine (4-5mg/kg) + 1/200,000 epinephrine was spraged into the abdominal cavity.
  Interventions: Drug: saline + intraperitoneal lidocaine
- Group IVPL(Intravenous and Intraperitoneal spray of lidocaine Group) (Experimental): At the beginning of the operation, intravenous infusion of reifentanil 0.1~0.2μg/kg/min, propofol 2~4mg/kg/h, rocuronium 0.3mg/kg/h intermittently, inhalation of 1%~2% sevoflurane were maintained, the fluctuation of blood pressure was not more than 20% of the basic level, and the heart rate was 50~100 times /min. 10 minutes before the infusion 2% lidocaine (1.5mg/kg) was administered to the patient. Subsequnetly, a continuous intravenous infusion 2% lidocaine ( 2mg/kg/h) was maintained until the end of the sugery. Before closing the abdominal cavity, 2% lidocaine (4-5mg/kg) + 1/200,000 epinephrine was spraged into the abdominal cavity.
  Interventions: Drug: intravenous + intraperitoneal lidocaine

INTERVENTIONS:
Drug: Saline — 10 minutes before the infusion saline 1.5mg/kg was administered to the patient. Subsequnetly, a continuous intravenous infusion saline 2mg/kg/h was maintained until the end of the sugery. Before closing the abdominal cavity, 20ml normal saline was administered.
  Other Names: placebo
  Arms: Group C(Control Group)
Drug: intravenous +saline lidocaine — 10 minutes before the infusion 2% lidocaine 1.5mg/kg was administered to the patient. Subsequnetly, a continuous intravenous infusion 2% lidocaine 2mg/kg/h was maintained until the end of the sugery. Before closing the abdominal cavity, 20ml normal saline was administered.
  Other Names: analgesic
  Arms: Group IV(Intravenous injection of lidocaine Group)
Drug: saline + intraperitoneal lidocaine — 10 minutes before the infusion saline 1.5mg/kg was administered to the patient. Subsequnetly, a continuous intravenous infusion saline ( 2mg/kg/h) was maintained until the end of the sugery. Before closing the abdominal cavity, 2% lidocaine (4-5mg/kg) + 1/200,000 epinephrine was spraged into the abdominal cavity.
  Other Names: intraperitoneal spary of lidocaine
  Arms: Group IP(Intraperitoneal spray of lidocaine Group)
Drug: intravenous + intraperitoneal lidocaine — 10 minutes before the infusion 2% lidocaine (1.5mg/kg) was administered to the patient. Subsequnetly, a continuous intravenous infusion 2% lidocaine ( 2mg/kg/h) was maintained until the end of the sugery. Before closing the abdominal cavity, 2% lidocaine (4-5mg/kg) + 1/200,000 epinephrine was spraged into the abdominal cavity.
  Other Names: intravenous and intraperitoneal injection of lidocaine
  Arms: Group IVPL(Intravenous and Intraperitoneal spray of lidocaine Group)

SUMMARY:
The purpose of this study is to determine whether laparoscopic spraying combined with intravenous injection of lidocaine can improve pain in patients undergoing laparoscopic myomectomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-65 years old;
2. ASA physical status classification I - III;
3. Undergoing laparoscopic hysteromyoma resection under general anesthesia;
4. The patient has been informed and has signed the informed consent form.

Exclusion Criteria:

1. Surgery duration exceeding 3 hours;
2. Need for additional surgery;
3. Allergy to the study drugs;
4. Presence of severe psychological,hepatic,renal,and cardiac diseases;
5. History of chronic pain or arrhythmia.

Elimination Criteria:

1. The patient or their family withdraws from or refuses to participate in the trial during the observation period;
2. Conversion from laparoscopy to laparotomy or change in surgical approach during the procedure.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of moderate to severe pain within 24 hours | Within 24 hours after surgery
  Pain severity was measured using The NRS((Numerical Rating Scale),The NRS≥4 was considered moderate to severe pain. If the NRS score is greater than or equal to 4 at least once within 24 hours, it is considered moderate to severe pain.

SECONDARY OUTCOMES:
NRS scores at different time intervals | 2 hours, 4 hours, 8 hours, 12 hours, 24 hours after surgery
  The severity of pain was measured using the NRS(Numerical Rating Scale), with NRS≥4 indicating moderate to severe pain. The NRS scores for movement, rest, and wound pain at 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours after surgery were observed to determine whether intraperitoneal spray combined with intravenous lidocaine could reduce the incidence of moderate to severe pain in patients undergoing laparoscopic myomectomy.
Sleep quality | Within 48h hours after surgery
  The subjective sleep status of Day 0, Day 1 and Day 2 was assessed using the AIS scale. For patients with an AIS score of 4 or higher, the Insomnia Severity Index (ISI) was used to classify the degree of insomnia.
Recovery quality | The first two days after surgery
  The Qor-15 scale was used to evaluate the recovery quality of patients in the first two days. QoR-15 Assessment Questionnaire:It includes five dimensions:physical comfort(5 items),physical independence(2 items),emotional state(4 items),psychological support(2 items),and pain(2 items). Scoring details: Each item is scored on an 11-point scale.Higher scores for positive items indicate higher frequency. The total score ranges from 0(worst recovery)to 150(best recovery).
The consumption of analgesic drugs. | Within 24 hours after surgery
  The consumption of analgesic drugs was recorded, defined as the cumulative consumption of opioids during surgery and the number and type of rescue medications used after surgery.
The number of lidocaine adverse reactions, postoperative nausea and vomiting, and the use of vasoactive drugs. | During surgery and within 24 hours after surgery
  The number of adverse reactions to lidocaine in patients during and within 24 hours after surgery was recorded, including tinnitus, perioral numbness, nystagmus, impaired consciousness, muscle twitching, convulsions, coma, bradycardia, arrhythmia, conduction block, hypotension, and circulatory collapse.
  The number and dosage of vasoactive drugs used by patients during surgery were recorded.
  The number of postoperative nausea and vomiting occurrences was recorded, defined as the recording of any nausea or vomiting within 24 hours after surgery.
BIS value | During the operation
  The BIS values of patients before surgery, before skin incision, 30 minutes into the surgery, and at the end of the surgery were recorded.
The time for recovery of bowel function | After surgery
  Record the recovery time of gastrointestinal function,which is defined as the time of the patient's first flatus,first defecation,and removal of the urinary catheter immediately after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China